CLINICAL TRIAL: NCT05420714
Title: Piloting the Use of Professional Continuous Glucose Monitoring at the Parkland Diabetes Clinic
Brief Title: Professional Continuous Glucose Monitoring at the Parkland Diabetes Clinic
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in study design to quality improvement
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Felona Gunawan, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STU-2021-1012
Record Dates: First submitted 2022-06-11; First posted 2022-06-15 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Diabete Mellitus
Keywords: continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Professional CGM Trial (Experimental): Participants will be asked to wear Dexcom Professional Continuous Glucose Monitoring (Pro-CGM) Device for 10 days. They will have 2 clinic visits with a certified diabetes care and education specialist (CDCES): initial visit for placement of the Pro-CGM and final visit to review the data with CDCES and their diabetes clinic provider. They will be asked to complete a short survey at the end of the 10 days about their experience using the Pro-CGM device and how it impacts their diabetes self-care practices.
  Interventions: Device: Dexcom Professional Continuous Glucose Monitoring

INTERVENTIONS:
Device: Dexcom Professional Continuous Glucose Monitoring — Patient will be asked to wear the Dexcom Pro-CGM device (small device that can be applied to either the arm or abdomen) for 10 days. They will have 30 minutes initial visit with CDCES to apply the device and review its use and 60 minute final session to review the blood sugar data from the CGM with CDCES and diabetes clinic provider.

SUMMARY:
The purpose of this study is to assess whether the short-term use of professional continuous glucose monitoring (Pro-CGM) at the Parkland Diabetes Clinic in selected patients with poorly-controlled diabetes due to hyper- and/or hypoglycemia leads to improvements in patients' glycemic control within 3-6 months, subjective understanding of how food, activity, and medications affect blood sugar levels, and diabetes self-care practices. The study will be a prospective cohort study that assesses patients glycemic control and diabetes self-care practices before and 3-6 months after utilization of a Pro-CGM for 10 days. Glycemic control and diabetes self-care practices will be assessed based on hemoglobin A1c measurements and glucose data download from glucometer and Pro-CGM. A short survey will be administered at the end of the 10 days Pro-CGM use to assess whether the Pro-CGM use had a positive impact on patients' understanding of how different activities affect their blood sugar and diabetes self-care practices.

Parkland Diabetes Clinic serves an ethnically diverse, low socioeconomic patient population, the majority of whom do not have access to diabetes technology like continuous glucose monitoring. CGM measures sugar levels every 5 to 15 minutes and have been shown in clinical studies to improve glycemic control. Establishing a professional CGM program at the clinic will provide short-term access to this technology. One of the main reason for conducting this study is to determine if Pro-CGM would be a useful intervention to integrate into the clinic's routine practice in the future.

ELIGIBILITY:
Inclusion Criteria:

Patients of the Parkland Diabetes Clinic who meets one or more of the following criteria:

* Patients with inaccurate HgbA1c due to conditions that affect red blood cell turnover (examples include but not limited to: anemia, hemoglobinopathies, chronic kidney disease)
* Patients with suspected recurrent hypoglycemia and/or hypoglycemia unawareness
* Patients with persistently elevated HgbA1c >8% despite reported adherence to medications and lifestyle modifications and after assessment by a Certified Diabetes Care and Education Specialist (CDCES)
* Patients with inability to do frequent fingersticks for blood glucose checks due to physical limitations (examples include but not limited to: vision loss, dexterity problems)

Exclusion Criteria:

* Patients who already have their own personal continuous glucose monitoring device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Average change in glycemic control 3 months after Pro-CGM use | 3 months
  Glycemic control will be assessed at baseline and 3 months after intervention by measuring hemoglobin A1c and/or obtaining 14-day average glucose from glucometer or CGM blood sugar data download. These data are collected as part of routine diabetes care at the clinic and will be obtained by chart review.

SECONDARY OUTCOMES:
Average change in hypoglycemia frequency 3 months after Pro-CGM use | 3 months
  Hypoglycemia frequency will be assessed at baseline and 3 months after intervention by reviewing 14-day fingerstick glucose data from glucometer download and comparing the % of blood sugar reading <70 mg/dL at baseline and 3 months after intervention. These data are collected as part of routine diabetes care at the clinic and will be obtained by chart review.
Average change in hyperglycemia frequency 3 months after Pro-CGM use | 3 months
  Hyperglycemia frequency will be assessed at baseline and 3 months after intervention by reviewing 14-day fingerstick glucose data from glucometer download and comparing the % of blood sugar reading >180 mg/dL at baseline and 3 months after intervention. These data are collected as part of routine diabetes care at the clinic and will be obtained by chart review.
Average change in frequency of fingerstick blood glucose checks 3 months after Pro-CGM use | 3 months
  The frequency of fingerstick glucose checks per day will be obtained from glucometer data download, which provides the average # of blood sugar reading per day, at baseline and 3 months after intervention. These data are collected as part of routine diabetes care at the clinic and will be obtained by chart review.
Percentage of positive patient response to the Pro-CGM Questionnaire | The survey will be administered at the end of the 10 days Pro-CGM use. The percentage of positive responses will be calculated at the end of study.
  The patients are given a questionnaire with 8 "Yes or No" questions about whether or not wearing the CGM has a positive impact on their diabetes self-care practices (diet, exercise, medication adherence, blood glucose monitoring). The percentage of "Yes" responses for the 8 questions will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Felona Gunawan, MD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey TS, Zisser HC, Garg SK. Reduction in hemoglobin A1C with real-time continuous glucose monitoring: results from a 12-week observational study. Diabetes Technol Ther. 2007 Jun;9(3):203-10. doi: 10.1089/dia.2007.0205. PMID 17561790
- [Background] Leinung M, Nardacci E, Patel N, Bettadahalli S, Paika K, Thompson S. Benefits of short-term professional continuous glucose monitoring in clinical practice. Diabetes Technol Ther. 2013 Sep;15(9):744-7. doi: 10.1089/dia.2013.0027. Epub 2013 Jun 20. PMID 23786229
- [Background] Kesavadev J, Vigersky R, Shin J, Pillai PBS, Shankar A, Sanal G, Krishnan G, Jothydev S. Assessing the Therapeutic Utility of Professional Continuous Glucose Monitoring in Type 2 Diabetes Across Various Therapies: A Retrospective Evaluation. Adv Ther. 2017 Aug;34(8):1918-1927. doi: 10.1007/s12325-017-0576-x. Epub 2017 Jun 30. PMID 28667580